CLINICAL TRIAL: NCT01773850
Title: Comparison of Carbon Nanotube X-ray Stationary Digital Breast Tomosynthesis and 2-D Digital Mammography in Patients With Known Breast Lesions.
Brief Title: Comparison of Stationary Breast Tomosynthesis and 2-D Digital Mammography in Patients With Known Breast Lesions
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC-1232
Record Dates: First submitted 2013-01-04; First posted 2013-01-23 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2017-04

CONDITIONS: Breast Neoplasms
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with a breast lesion undergoing surgical biopsy. All patients will undergo stationary Carbon Nanotube x-ray digital breast tomosynthesis imaging in addition to routine conventional digital mammography.
  Interventions: Device: Stationary Carbon Nanotube X-ray Digital Breast Tomosynthesis Scanner

INTERVENTIONS:
Device: Stationary Carbon Nanotube X-ray Digital Breast Tomosynthesis Scanner — All patients will undergo conventional imaging and imaging with the carbon nanotube based x-ray stationary digital breast tomosynthesis scanner device.
  Other Names: Carbon nanotube based x-ray digital breast tomosynthesis (CNT SDBT) Scanner

SUMMARY:
The goal of the study is to compare the radiologist confidence level in evaluating patients with known breast lesions using a carbon nanotube x-ray based stationary breast tomosynthesis imaging device. The comparison will be made against conventional mammography acquired as a part of a standard clinical workup. One hundred patients who are to have a clinical surgical breast biopsy will be recruited for the study. A reader study will be performed to evaluate the ROC characteristics of the system.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years old.
* Scheduled for breast biopsy of at least one breast lesion.
* Lesion detected on mammogram.
* Symptomatic by patient self-report, patient self-breast exam or clinical exam.
* Able to provide informed consent.

Exclusion Criteria:

* Male. (It is uncommon for men to present for imaging and the overwhelming majority of findings are non-cancerous and do not lead to biopsy; male breast cancer represents <1% of newly diagnosed breast cancer)
* Less than 18 years of age.
* Patient unable to give consent.
* Institutionalized subject (prisoner or nursing home patient).
* Any woman who is pregnant or has reason to believe she is pregnant or any woman who is lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical breast biopsies for lesions detected on mammograms.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Receiver Operative Curve (ROC) Area Under the Curve (AUC) (percentage) | approximately 18 months
  Receiver Operative Curve (ROC) Area Under the Curve (AUC) analysis of the stationary breast tomosynthesis (SDBT) system for the the characterization of suspicious breast lesions in comparison to x-ray mammography.

SECONDARY OUTCOMES:
Reader preference - arbitrary units | approximately 18 months
  To evaluate radiologists confidence in evaluating specific lesion characteristics in suspicious breast lesions. Readers will be scored from -3 to +3.

CONTACTS AND LOCATIONS:
Overall Officials: Yueh Z Lee, MD,PhD, Principal Investigator — University of North Carolina, Chapel Hill; Cherie M Kuzmiak, DO, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Qian X, Tucker A, Gidcumb E, Shan J, Yang G, Calderon-Colon X, Sultana S, Lu J, Zhou O, Spronk D, Sprenger F, Zhang Y, Kennedy D, Farbizio T, Jing Z. High resolution stationary digital breast tomosynthesis using distributed carbon nanotube x-ray source array. Med Phys. 2012 Apr;39(4):2090-9. doi: 10.1118/1.3694667. PMID 22482630